CLINICAL TRIAL: NCT04489589
Title: Midodrine for the Early Liberation of Vasopressor Support in the ICU - The LIBERATE Pilot Study
Brief Title: Midodrine for the Early Liberation of Vasopressor Support in the ICU
Acronym: LIBERATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other); Institute of Health Economics, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00096716
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Shock
MeSH Terms: conditions — Critical Illness; Shock | interventions — Midodrine; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midodrine (Experimental): Midodrine 10mg PO/NG q8h
  Interventions: Drug: Midodrine
- Placebo (Placebo Comparator): Microcrystalline cellulose PO/NG q8h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine — 10mg PO/NG q8h
  Other Names: Midodrine Hydrochloride
  Arms: Midodrine
Drug: Placebo — 10mg PO/NG q8h
  Other Names: Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Vasopressors are medications that are given intravenously to increase the blood pressure of patients with illnesses that cause dangerous blood pressure drops. When a doctor prescribes a vasopressor, they ask that the dose be adjusted to achieve a specific blood pressure. This kind of medical support with intravenous (IV) vasopressors are usual treatments in intensive care unit (ICU) settings. Oral vasopressors, such as midodrine, have been historically used to maintain blood pressure in non-critically ill patients. In this study, the investigators will be using midodrine to reduce the need for IV vasopressors as blood pressure improves during the stay in the ICU

The LIBERATE pilot study will evaluate the role of midodrine for patients with low blood pressure in the ICU. The investigators are planning on enrolling up to 20 study participants to evaluate this question in the General Systems ICU at the University of Alberta Hospital.

DETAILED DESCRIPTION:
Purpose: Resuscitation and hemodynamic support with intravenous (IV) vasopressors is a prime indication of treatment in intensive care unit (ICU) settings. Hemodynamic support is typically provided with intravenous (IV) vasopressors. However, these have been shown to have significant negative effects including increased central venous catheter line associated infections, venous thromboembolic disease, impaired mobility and gastrointestinal injury and ischemia. Oral vasopressors, such as midodrine, have been historically used for hemodynamic support in non-critically ill patients, but their study in patients as IV pressor sparing therapy has been limited.

Hypothesis: to evaluate the expanded role of midodrine for any vasoplegic patients in the ICU.

Justification: In 2018, there were 1,613 admissions to the adult general systems ICU (GSICU) at the University of Alberta Hospital (UAH). Patients were sick, with a mean Acute Physiology and Chronic Health Evaluation II (APACHE) score of 21.3, with 36.4% requiring vasopressors on admission, accounting for 1942 patient-days (data from eCritical TRACER database). In the environment strained healthcare resources and limited ICU capacity, the ability to safely wean patients from IV vasopressors with transition to oral hemodynamic supporting agents would greatly improve how patients navigate through the healthcare system. This in turn will improve patient-centered case.

Primary Objective:

To determine if recruitment for LIBERATE is achievable and feasible To compare the effect of enteral midodrine vs placebo on duration of vasopressor support

Secondary Objective: To compare the effect of enteral midodrine vs. placebo on:

ICU length of stay 90-day all-cause mortality Rate of re-initiation of IV vasopressors Rates of ICU re-admission Adverse events Research Method/Procedures: The LIBERATE Trial is a single centre, concealed-allocation parallel-group blinded pilot RCT. Patients will be randomly assigned to midodrine (enteral, 10mg every 8h) or placebo (microcrystalline cellulose) for the duration of their IV vasopressor therapy and 24h following the discontinuation of their IV vasopressor therapy. The recruitment target is 60 patients (i.e., 30 patients per arm) with full follow-up to ensure feasibility. Study personnel at the clinical sites will document the ICU length of stay. Daily assessment will occur for re-initiation of IV vasopressors and ICU re-admission. Patients will be followed at 90 days for mortality.

Plan for Data Analysis: Analyses of the primary and secondary outcomes will involve summary measures obtained by aggregating the endpoints using Stata software package (StataCorp, Texas, USA). Baseline comparisons will be performed using chi-squared test for equal proportions with results to be reported as numbers, percentages, and 95% confidence intervals. Continuous normally distributed variables will be compared using paired t-tests and reported as means with 95% confidence intervals, while non-normally distributed will be compared using Wilcoxon rank sum tests and reported as medians and interquartile ranges.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* ICU admission
* Ongoing vasopressor support
* Decreasing vasopressor dose

Exclusion Criteria:

* Greater than 24 hours from peak vasopressor dose
* Contraindication to enteral medications
* Previously on midodrine in last 7 days
* Expected death or withdrawal of life-sustaining therapies
* Pregnancy
* Known allergy to Midodrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Rates | 1 year
  Recruitment metrics by patients recruitment and consent rate
Duration of vasopressor support | 1 year
  Duration of intravenous vasopressor support

SECONDARY OUTCOMES:
ICU length of stay | 1 year
  Total duration of patient stay in ICU
Mortality | Up to 90 days
  All cause patient mortality within 90 days of study recruitment
Re-initiation of IV vasopressors | 1 year
  Rate of re-initiation of intravenous vasopressors during ICU stay
ICU re-admissions | 1 year
  Rates of ICU re-admissions during same hospitalization
Adverse events | 1 year
  Rates of adverse events during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Oleksa G Rewa, MD MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, all results will be used to inform the development of a larger scale, multi centre RCT.

REFERENCES:
- [Derived] Kilcommons SJ, Hammal F, Opgenorth DL, Fiest KM, Karvellas CJ, Lau VI, MacIntyre E, Senaratne J, Slemko J, Sligl W, Zampieri F, Duquette D', Guan LT, Baig N, Bagshaw SM, Rewa OG. Midodrine for the early liberation from vasopressor support in the ICU (LIBERATE): a feasibility study. Pilot Feasibility Stud. 2024 Dec 4;10(1):147. doi: 10.1186/s40814-024-01577-2. PMID 39633467